CLINICAL TRIAL: NCT02245906
Title: Investigation on Effect of Brazilian Fruits on Glucose and Insulin Responses, Anti-inflammatory Properties, Antioxidative Capacity and Satiety in Healthy Subjects
Brief Title: Effect of Brazilian Fruits Peel on Metabolic Regulation and Appetite in Healthy Subjects
Acronym: BRASIL-MET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Elin Östman, Assoc. Prof, PhD, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BRASIL-MET
Record Dates: First submitted 2014-09-16; First posted 2014-09-22 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: Brazilian fruit peel; Functional food; Cardiometabolic risk; Metabolic syndrome; Inflammation; Appetite; Gut hormone
MeSH Terms: conditions — Metabolic Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control drink (Placebo Comparator): 300 ml control drink containing equal amount of total fiber and pectine as Brazilian fruit drink, acute study / one time administration
  Interventions: Dietary Supplement: Control drink
- Brazilian fruit peel (Experimental): 300 ml test drink containing Brazilian fruit peel flour, acute study / one time administration
  Interventions: Dietary Supplement: Brazilian fruit peel flour
- Negative control drink (Placebo Comparator): 300 ml control drink without containing amount of total fiber and pectine as Brazilian fruit drink, acute study / one time administration
  Interventions: Dietary Supplement: Negative control drink

INTERVENTIONS:
Dietary Supplement: Control drink — As a control, subjects are asked to consume 300 ml control drinks containing equal amount of total fiber and pectine as Brazilian fruit drink. Following 10 min. beverage consumption, subjects will be given standardized breakfast corresponding to 50 g carbohydrate.
  Arms: Control drink
Dietary Supplement: Brazilian fruit peel flour — In this study, subjects are asked to consume 300 ml beverage drinks contain certain amounts of Brazilian fruit peel flour. Following 10 min. beverage consumption, subjects will be given standardized breakfast corresponding to 50 g carbohydrate.
  Arms: Brazilian fruit peel
Dietary Supplement: Negative control drink — As a negative control, subjects are asked to consume 300 ml control drinks without containing amount of total fiber and pectine as Brazilian fruit drink. Following 10 min. beverage consumption, subjects will be given standardized breakfast corresponding to 50 g carbohydrate.
  Arms: Negative control drink

SUMMARY:
The purpose of the study was to investigate how Brazilian fruits peel affect acute/postprandial glucose and insulin responses, inflammatory markers, appetite control peptides, antioxidative capacity, as well as subjective appetite ratings (VAS-visual analogue scales) in healthy volunteers. We hypothesize that certain Brazilian fruits peel added to a standardized meal will improve postprandial glucose tolerance and other metabolic biomarkers in healthy volunteers, compared with a similar meal without the corresponding plant materials.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Signed informed consent
* BMI 20 - 28 kg/m2 with weight change <3 kg latest 2 months
* Must be able to accept plant-based foods/drinks

Exclusion Criteria:

* Below 18 years
* Uncomfortable speaking English and/or difficulties in understanding spoken English
* Smoking or using snuff
* Vegetarian or vegan
* Stressed by venous blood sampling or previous experience of being difficult to cannulate
* Receiving any drug treatment that may influence the study outcomes
* Pregnancy or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changing on blood glucose concentration after treatment with brazilian fruits peel | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 min
  The capillary blood samples will be taken for blood glucose analysis

SECONDARY OUTCOMES:
Changing on subjective appetite ratings after treatment with Brazilian fruits peel | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 min.
  Appetite will be assessed using standard subjective 100 mm VAS (visual analogue scale) at time intervals throughout each visit
Identify plasma metabolite profile (untargeted approach) after treatment with Brazilian fruits peel | Prior to the initial intervention at 0 min and after intervention at 60, 90, 120, 180 min.
  Metabolite profile will be analyzed using Liquid Chromatography-Mass Spectrometry based methods
Changing on insulin after treatment with Brazilian fruits peel | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 min.
  The venous serum blood samples will be taken for insulin analysis
Changing on inflammatory markers (i.e. interleukin-6, interleukin-8, tumor necrosis factor-alpha, necrosis factor kappa-beta, adiponectin and C-reactive protein) after treatment with Brazilian fruits peel | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 min.
  The venous serum blood samples will be taken for inflammatory markers analysis
Changing on appetite markers (i.e. ghrelin, cholecystokinin, glucagon-like peptide-1, gastric inhibitory polypeptide, peptide YY, amylin, pancreatic polypeptide) after treatment with Brazilian fruits peel | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 min.
  The venous serum blood samples will be taken for appetite markers analysis

CONTACTS AND LOCATIONS:
Overall Officials: Elin Östman, PhD, Principal Investigator — Lund University; Glaucia Lima, MSc, Study Chair — Lund University; Yoghatama Cindya Zanzer, MSc, Study Chair — Lund University
Locations (1):
- Antidiabetic Food Centre (Medicon Village) - Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No